CLINICAL TRIAL: NCT04501588
Title: Parent Language Intervention for Autism
Brief Title: Parent Telehealth Intervention for Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Megan Roberts, Associate Professor of Communication Sciences and Disorders, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00201708
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: autism; parent intervention; parent coaching; early intervention; parent-mediated intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Children will enroll in the study between 18-48 months of age and will be randomly assigned to either receive responsive training with video feedback or responsive training without video feedback.
Who Masked: Outcomes Assessor
Masking Description: Assessors who score/code the parent-child interaction are blind to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parent Learning Style 1 (Experimental): Mothers with Learning Style 1 will be randomly assigned to receive the responsive intervention with video feedback or without video feedback.
  Interventions: Behavioral: Responsive training with no video feedback
- Parent Learning Style 2 (Experimental): Mothers with Learning Style 2 will be randomly assigned to receive the responsive intervention with video feedback or without video feedback.
  Interventions: Behavioral: Responsive training with video feedback
- Learning Style 1 (Parent) (Active Comparator): Mothers with Learning Style 1 will be randomly assigned to receive the responsive intervention with video feedback or without video feedback.
  Interventions: Behavioral: Responsive training with video feedback
- Learning Style 2 (Parent) (Active Comparator): Mothers with Learning Style 2 will be randomly assigned to receive the responsive intervention with video feedback or without video feedback.
  Interventions: Behavioral: Responsive training with no video feedback

INTERVENTIONS:
Behavioral: Responsive training with no video feedback — Parents will receive responsive training, but will not watch themselves on video to reflect on their strategy use.
  Other Names: No Video Feedback
  Arms: Learning Style 2 (Parent); Parent Learning Style 1
Behavioral: Responsive training with video feedback — Parents will receive responsive training and watch themselves on video to reflect on their strategy use.
  Other Names: Video Feedback
  Arms: Learning Style 1 (Parent); Parent Learning Style 2

SUMMARY:
As a result of the COVID-19 pandemic, telecoaching/telepractice models are of urgent importance. Given this, parents in the study will receive parent coaching through weekly video calls. To help us understand the best types of telecoaching, we will offer all participants responsive coaching, with half of the participants receiving an additional opportunity to reflect on their own use of language strategies with a therapist using video feedback and the other half receiving responsive coaching as usual, without video feedback. This information is important in helping us to understand the best way to coach parents using a telepractice model so that parents implement the intervention at high fidelity. Furthermore, we will aim to understand how parent learning style may also influence the implementation of these strategies.

ELIGIBILITY:
Inclusion Criteria:

Child inclusion criteria include:

* diagnosis of ASD or showing signs of ASD based on autism screening
* chronological age of less than 48 months
* a parent who is willing to learn intervention strategies
* English as the primary language spoken in the home

Parent inclusion criteria include:

- Biological Mother

Exclusion Criteria:

* Children or parents with additional impairments (e.g., blindness, deafness, genetic syndromes) will be excluded from the study.
* Fathers or caregivers other than the child's Mother will be excluded from the study.

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Parent Use of Language Support Strategies (Mother-child interaction) | Two months after the start of the study
  Mother use of intervention strategies will be measured by transcribing and coding mother behaviors during 12-minute parent-child interactions, using a standard set of toys. The primary dependent variable will be the amount of correct strategy used expressed as a percentage correct. This is the percentage of child communication to which the adult responds correctly (i.e., contingently and within 5 seconds).

SECONDARY OUTCOMES:
MacArthur-Bates Communicative Development Inventory (MCDI) (Child) | Two months after the start of the study
  Parent report of child's expressive vocabulary and prelinguistic communication skills

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
N/A at this time

REFERENCES:
- [Background] Roberts MY, Kaiser AP. Early intervention for toddlers with language delays: a randomized controlled trial. Pediatrics. 2015 Apr;135(4):686-93. doi: 10.1542/peds.2014-2134. Epub 2015 Mar 2. PMID 25733749

DOCUMENTS (1):
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT04501588/ICF_000.pdf